CLINICAL TRIAL: NCT07014267
Title: Virtual Reality for Mindfulness and Anxiety Reduction in Fertility Procedures
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ART Fertility Clinics LLC (Other)
Responsible Party: Principal Investigator, Laura Melado, Medical Director - Abu Dhabi, ART Fertility Clinics LLC
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2503-ABU-007-LMV
Record Dates: First submitted 2025-03-20; First posted 2025-06-10 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-05

CONDITIONS: Virtual Reality; Patient Experience
Keywords: anxiety; stress; pain perception; recovery duration; virtual reality
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No VR intervention) (No Intervention): Patients will receive standard care without the VR intervention. Anxiety levels will be measured using the State-Trait Anxiety Inventory (STAI) before the procedure (baseline) and after the procedure.
- Intervention Group (Virtual Reality Intervention) (Experimental): Patients will experience the VR mindfulness intervention using the Tripp App or comparable applications.
  Anxiety levels will be measured using the STAI before the VR experience, immediately after the VR experience, and after the procedure.
  Interventions: Device: Intervention Group (Virtual Reality intervention)

INTERVENTIONS:
Device: Intervention Group (Virtual Reality intervention) — Patients will experience the VR mindfulness intervention using the Tripp App or comparable applications.
  Anxiety levels will be measured using the STAI before the VR experience, immediately after the VR experience, and after the procedure.
  Arms: Intervention Group (Virtual Reality Intervention)

SUMMARY:
This study aims to evaluate the effectiveness of a Virtual Reality (VR)-based mindfulness and meditation intervention in reducing anxiety among patients undergoing fertility-related surgical procedures. Anxiety is a common challenge in fertility treatments, often leading to emotional distress and increased pain perception. By incorporating a non-invasive VR intervention, the investigators seek to improve patient experience, minimize preoperative anxiety, and potentially reduce postoperative discomfort and recovery times. This randomized controlled trial (RCT) will compare standard care with a VR intervention in a clinical setting, measuring key outcomes such as anxiety levels, pain perception, recovery duration, and overall patient satisfaction. The findings may contribute to more patient centered fertility care, offering an innovative, scalable, and cost-effective approach to anxiety management in reproductive medicine.

DETAILED DESCRIPTION:
This study examines the effectiveness of a Virtual Reality (VR) mindfulness intervention in reducing anxiety for patients undergoing fertility surgeries. The trial will compare VR with standard care, measuring outcomes like anxiety, pain, recovery time, and patient satisfaction. The results could provide a cost-effective, patient-centered approach to managing anxiety in fertility treatments.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-50.
* Scheduled for fertility-related surgical procedures.
* Able to provide informed consent.

Exclusion Criteria:

* History of motion sickness or VR-related discomfort.
* Cognitive or psychological conditions affecting participation.
* Procedures requiring emergency intervention.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 500 (Estimated)
Dates: Start 2025-07-10 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in anxiety level before and after the intervention | 10 minutes before the procedure and 10 minutes after procedure (intervention group and control group)
  Measured using the State-Trait Anxiety Inventory (STAI), which provides a score from 20 to 80. Higher scores indicate more anxiety. Change from baseline to post-procedure will be compared between VR and control groups. Score on STAI (range 20-80)

SECONDARY OUTCOMES:
Visual Facial Anxiety Scale Score | 10 minutes before the procedure and 10 minutes after procedure (intervention group and control group)
  A 6-tier visual facial anxiety scale used to assess preoperative anxiety. Scores range from 1 (most anxious) to 6 (least anxious). Will be used as an alternative assessment alongside STAI. Visual scale score (1-6)
Pain Score | Immediately post-procedure
  Pain levels will be assessed using a 10-point Numeric Rating Scale (NRS). Higher scores indicate greater pain. NRS score (0-10)
Amount of Pain Medication Used | During and immediately after procedure
  Total amount of analgesics or anesthetics administered, based on patient record and clinical protocol (measured in mg)
Recovery Time | 30 minutes after the end of procedure (before discharge).
  Measured in minutes to determine the duration of post-operative recovery.
Composite Patient Satisfaction Score | 30 minutes after the end of procedure (before discharge).
  10-item emoji-based questionnaire scored from 1-5 or 1-3 per item, depending on the scale used. Total composite score ranges from 10-50 or 10-30. Higher scores indicate greater satisfaction. May be normalized to 0-100%. Unites of measure: Composite score (10-50) or percentage (0-100%)
Recovery Time | 30 minutes after the end of procedure (before discharge).
  Duration of patient recovery (minutes)
Gender-specific Effectiveness | Through study completion, an average of 1 year
  Subgroup analysis of anxiety reduction by gender (male vs. female). Measured using the State-Trait Anxiety Inventory (STAI), which provides a score from 20 to 80. Higher scores indicate more anxiety. Change from baseline to post-procedure will be compared between VR and control groups. Score on STAI (range 20-80)
Procedure-specific Effectiveness | Through study completion, an average of 1 year
  Subgroup analysis of primary outcome by procedure type. Measured using the State-Trait Anxiety Inventory (STAI), which provides a score from 20 to 80. Higher scores indicate more anxiety. Change from baseline to post-procedure will be compared between VR and control groups. Score on STAI (range 20-80). Difference in mean STAI score change by procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Lawrenz, Research Director, Study Director — ART Fertility Clinics LLC
Locations (1):
- ART Fertility Clinics LLC, Abu Dhabi, United Arab Emirates

IPD SHARING:
Plan to Share IPD: Undecided
upon request